CLINICAL TRIAL: NCT04509648
Title: One-week Hypofractionated Radiotherapy in Breast Cancer Patients With an Indication for Regional Nodal Irradiation: Prospective, Single-arm Trial
Brief Title: Adjuvant Regional Nodal Radiation Therapy for One Week in Breast Cancer
Acronym: ARROW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, CAOLU, Associated professor of Department of Radiation Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC-SHF RNI
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: regional nodal irradiation; IMRT; IMPT; internal mammary nodes irradiation; Super Hypofractionated irradiation to tumor bed boost; Super Hypofractionated irradiation for one week
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Super Hypofractionated radiotherapy (Experimental): Patients with an indication for regional nodal irradiation will receive 5.2 Gy in 5 fractions to chest wall or whole breast and regional lymph regions (including supraclavicular/infraclavicular region, internal mammary nodes, and any part of the axillary bed at risk) and a sequential tumor bed boost of 5.2 Gy in 2 fractions to the conserved breast at the discretion of radiation oncologist.
  Interventions: Radiation: External Beam radiotherapy using IMRT technique

INTERVENTIONS:
Radiation: External Beam radiotherapy using IMRT technique — 2600cGy/ 5 fractions / 1 weeks to ipsilateral chest wall or whole breast and regional lymph regions and a sequential tumor bed boost of 5.2 Gy in 2 fractions to the conserved breast

SUMMARY:
The purpose of this trial is to investigate the toxicities and efficacy of super hypofractionated regional nodal radiotherapy (RNI) for one week in breast cancer patients treated with mastectomy or breast conserving surgery. Super hypofractionated radiotherapy will be delivered to chest wall or whole breast and regional lymph regions (including supraclavicular/infraclavicular region, internal mammary nodes, and any part of the axillary bed at risk). Eligible breast cancer patients will be followed for at least 5 years to evaluate the acute and late radiation-induced toxicities, locoregional recurrence, over survival, distant metastasis, and quality of life.

DETAILED DESCRIPTION:
Eligible breast cancer patients will receive super hypofractionated radiotherapy of 5.2 Gy in 5 fractions within one week and a sequential tumor bed boost of 5.2 Gy in 2 fractions to the conserved breast. The dose is prescribed to ipsilateral chest wall or whole breast and regional lymph regions (including supraclavicular/infraclavicular region, internal mammary nodes, and any part of the axillary bed at risk). All patients are treated with intensity modulated radiation therapy (IMRT) technique or intensity modulated proton therapy (IMPT). The primary endpoint is ≥2 grade any acute radiation induced toxicity event. Patients will be followed for at least 5 years to evaluate the acute and late radiation-induced toxicity, locoregional recurrence, over survival, distant metastasis, and quality of life.

Calculation of the required number of cases based on an alpha of 0.05 and a power of 80% with a maximal tolerable toxicity difference of 10% during and within 6 months after RNI comparing to conventional radiotherapy and lost rate of follow up of 10%. In total 197 patients are needed to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old
* Pathologically invasive breast cancer
* Undergoing BCS or mastectomy with reconstruction allowed, along with axillary lymph node dissection or sentinel lymph node biopsy.
* Axillary lymph node metastasis confirmed histologically (involving one or more nodes), or node-negative axilla with an indication for RNI as determined by the radiation oncologist.
* Karnofsky Performance Status scoring ≥80, and anticipative overall survival >5 years
* Surgery wound healed without infection
* Negative pathologically surgical margin
* Estrogen-receptor, Progesterone-receptor, HER-2, and Ki67 index assessment on the primary breast tumor or axillary nodes is feasible.
* Women of child-bearing potential must agree to use adequate contraception for up to 1 month before study treatment and the duration of study participation
* Ability to understand and willingness to participate the research and sign the consent forms

Exclusion Criteria:

* Pathologically positive ipsilateral supraclavicular lymph node
* Pathologically or radiologically confirmed involvement of ipsilateral internal mammary lymph nodes
* Pregnant or lactating women
* Severe non-neoplastic medical comorbidities that preclude radiation treatment (e.g., severe ischemic heart disease, arrhythmia, chronic obstructive pulmonary disease).
* History of non-breast malignancy within 5 years with the exception of lobular carcinoma in situ, basal cell carcinoma of the skin, carcinoma in situ of skin, Adenocarcinoma in situ of the lung and carcinoma in situ of the cervix
* simultaneous contralateral breast cancer or a prior history of ipsilateral breast cancer (including DCIS).
* Previous radiotherapy to the neck, chest and/or ipsilateral axillary region
* Active collagen vascular disease
* Definitive pathological or radiologic evidence of distant metastatic disease
* Primary T4 tumor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative complication rate of ≥Grade 2 Acute Radiation-induced Toxicity | 6 months
  Within time from the beginning of radiotherapy to 6 months after completion of radiotherapy, any acute radiation-induced toxicities will be assessed and recorded after the last fraction using the Common Terminology Criteria for Adverse Events (CTCAE) 3.0.

SECONDARY OUTCOMES:
Cumulative complication rate of ≥Grade 2 Late Radiation-induced Toxicity | 5 years
  Within time from 6 months after completion of radiotherapy to 5 years after completion of radiotherapy, any late toxicity will be assessed and recorded using the Radiation Therapy Oncology Group (RTOG) /European Organization for Research on Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring Schema and CTCAE 3.0
Number of Participants with excellent or good Cosmetic outcomes following breast conserving surgery-Harvard/ NSABP/RTOG scoring scale | 6 months
  The cosmetic outcomes will be evaluated at 6 months after last fractions. The cosmetic outcomes are evaluated based on the Allegheny General Modification of the Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/ RTOG scoring scale which graded patients into the following four classifications: excellent, when compared to the untreated breast, there is a minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast
Number of Participants with excellent or good Cosmetic outcomes following breast conserving surgery-Harvard/ NSABP/RTOG scoring scale | 5 years
  The cosmetic outcomes will be evaluated at 5 years after last fractions. The cosmetic outcomes are evaluated based on the Allegheny General Modification of the Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/ RTOG scoring scale which graded patients into the following four classifications: excellent, when compared to the untreated breast, there is a minimal or no difference in the size or shape of the treated breast; good, slight difference in the size or shape of the treated breast; fair, obvious difference in the size or shape of the treated breast; and poor, marked change in the size or shape of the treated breast
Locoregional recurrence | 5 years
  any first recurrence confirmed by histology or cytology within the ipsilateral chest wall and/or regional nodes area(including supraclavicular, infraclavicular or internal mammary lymph nodes)
Distant metastasis free survival (DMFS) | 5 years
  The time from the date of enrollment to any recurrence of tumor at distant sites or death from any cause
Invasive recurrence-free survival (IRFS) | 5 years
  The time from the date of enrollment to any invasive recurrence of tumor or death from any cause
Over survival (OS) | 5 years
  The time from the date of enrollment to the date of death from any cause

OTHER OUTCOMES:
Quality of Life-EORTC QLQ-C30 | 6 months
  Quality of life will be assessed before radiotherapy and 6 months after last fractions using self administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC BR-23 | 6 months
  Quality of life will be assessed before radiotherapy and 6 months after last fractions using self administered questionnaire EORTC QLQ-BR23
Quality of Life-EORTC QLQ-C30 | 5 years
  Quality of life will be assessed before radiotherapy and 5 years after last fractions using self administered questionnaire EORTC QLQ-C30
Quality of Life-EORTC BR-23 | 5 years
  Quality of life will be assessed before radiotherapy and 5 years after last fractions using self administered questionnaire EORTC QLQ-BR23

CONTACTS AND LOCATIONS:
Overall Officials: Lu Cao, PhD, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie J, Zheng S, Qi WX, Gan L, Yu B, Jiang J, Zhang J, Shi Y, Dong M, Cai G, Cai R, Xu C, Xu H, Qian X, Zhang Y, Chen M, Cao L, Chen J. One-week regimen for postoperative regional irradiation in breast cancer: the ARROW trial protocol. BMJ Open. 2025 May 15;15(5):e096677. doi: 10.1136/bmjopen-2024-096677. PMID 40379319